CLINICAL TRIAL: NCT06031688
Title: A Randomized Phase II Study of Tepotinib With or Without Ramucirumab in Participants With MET Exon 14 Skipping Positive Stage IV or Recurrent Non-Small Cell Lung Cancer (LUNG-MAP SUB-STUDY)
Brief Title: Targeted Treatment for Advanced Non-Small Cell Lung Cancer That Has a MET Exon 14 Skipping Gene Change (An Expanded Lung-MAP Treatment Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1900K; NCI-2023-04727 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1900K (Other: SWOG); S1900K (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Ramucirumab; tepotinib; EMD1214063

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: (Ramucirumab and tepotinib) (Experimental): Patients receive ramucirumab IV over 30-60 minutes on day 1 of each cycle and tepotinib PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients optionally undergo lymphoscintigraphy scan at screening prior to treatment, at the first occurrence of peripheral edema (defined as the development of grade ≥ 1 CTCAE Edema Limbs affecting either the arms, hands, or legs), and if peripheral edema increases in attribution. Patients also undergo blood collection, CT scan and/or MRI throughout the trial. Additionally, patients undergo urine collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Lymphoscintigraphy; Procedure: Magnetic Resonance Imaging; Biological: Ramucirumab; Drug: Tepotinib
- Arm B: (Tepotinib) (Active Comparator): Patients receive tepotinib PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients optionally undergo lymphoscintigraphy scan at screening prior to treatment, at the first occurrence of peripheral edema (defined as the development of grade ≥ 1 CTCAE Edema Limbs affecting either the arms, hands, or legs), and if peripheral edema increases in attribution. Patients also undergo blood collection, CT scan and/or MRI throughout the trial. Additionally, patients undergo urine collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Lymphoscintigraphy; Procedure: Magnetic Resonance Imaging; Drug: Tepotinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Lymphoscintigraphy — Undergo lymphoscintigraphy scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Ramucirumab — Given IV
  Other Names: Anti-VEGFR-2 Fully Human Monoclonal Antibody IMC-1121B; Cyramza; IMC 1121B; IMC-1121B; IMC1121B; LY 3009806; LY-3009806; LY3009806; Monoclonal Antibody HGS-ETR2
  Arms: Arm A: (Ramucirumab and tepotinib)
Drug: Tepotinib — Given PO
  Other Names: c-Met Inhibitor MSC2156119J; EMD 1214063; EMD-1214063; EMD1214063; MSC 2156119; MSC 2156119J; MSC-2156119; MSC-2156119J; MSC2156119; MSC2156119J

SUMMARY:
This phase II Expanded Lung-MAP treatment trial tests tepotinib with or without ramucirumab for the treatment of patients with advanced non-small cell lung cancer that has spread from where it first started (primary site) to other places in the body (stage IV) or that has come back after a period of improvement (recurrent). Tepotinib is used in patients whose cancer has a mutated (changed) form of a gene called MET. It is in a class of medications called kinase inhibitors. It works by blocking the action of the abnormal MET protein that signals tumor cells to multiply. This helps slow or stop the spread of tumor cells. Ramucirumab is a monoclonal antibody that may prevent the growth of new blood vessels that tumors need to grow. Giving tepotinib with ramucirumab may lower the chance of the cancer from growing or spreading in patients with stage IV or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the response rate (confirmed or unconfirmed, complete or partial) between participants with MET exon 14 skipping positive non-small cell lung cancer (NSCLC) randomized to tepotinib with or without ramucirumab.

SECONDARY OBJECTIVES:

I. To compare the frequency of all-grade treatment- related peripheral edema as defined by Common Terminology Criteria for Adverse Events (CTCAE) between the arms.

II. To evaluate the frequency and severity of toxicities within each arm. III. To compare progression-free survival between the arms. IV. To compare overall survival between the arms. V. To estimate the duration of response (DoR) among responders within each arm.

TRANSLATIONAL MEDICINE OBJECTIVE:

I. To establish a tissue/blood repository for participants with MET exon 14 skipping non-small cell lung cancer (NSCLC).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive ramucirumab intravenously (IV) over 30-60 minutes on day 1 of each cycle and tepotinib orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive tepotinib PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients optionally undergo lymphoscintigraphy scan at screening prior to treatment, at the first occurrence of peripheral edema (defined as the development of grade ≥ 1 CTCAE Edema Limbs affecting either the arms, hands, or legs), and if peripheral edema increases in attribution. Patients also undergo blood collection, computed tomography (CT) scan and/or magnetic resonance imaging (MRI) throughout the trial. Additionally, patients undergo urine collection during screening and on study.

After completion of study treatment, patients are followed-up every 12 weeks or more often as clinically indicated until progression and then every 6 months for 2 years and at the end of 3 years from date of sub-study randomization.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been assigned to S1900K by the Southwest Oncology Group (SWOG) Statistics and Data Management Center (SDMC). Assignment to S1900K is determined by the LUNGMAP protocol
* Participants must have documentation of stage IV or recurrent NSCLC with a MET exon 14 skipping mutation determined by tissue-based or blood-based (circulating tumor DNA [ctDNA]) next generation sequencing (NGS) assay done within a laboratory with Clinical Laboratory Improvement Act (CLIA), International Organization for Standardization (ISO)/ International Electrotechnical Commission (IEC), College of American Pathologists (CAP), or similar certification. Documentation must either be:

  * NGS test results from tissue submitted for LUNGMAP screening, or
  * Submitted documentation in the LUNGMAP Rave Electronic Data Capture System of a MET exon 14 skipping mutation from a previously completed tissue or blood-based NGS test
* Participants must have measurable disease documented by CT or MRI. The CT from a combined positron emission tomography (PET)/CT may be used to document measurable disease ONLY if it is of diagnostic quality, otherwise, it may be used to document non-measurable disease only. Measurable disease must be assessed within 28 days prior to sub-study randomization. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to sub-study randomization. All known sites of disease must be assessed and documented on the Baseline Tumor Assessment Form. Participants whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to sub-study randomization to be considered measurable
* Participants must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to sub-study randomization
* Participants must not have leptomeningeal disease, spinal cord compression or brain metastases unless:

  * Metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 3 days following the stereotactic radiation and/or 14 days following whole brain radiation, and prior to sub-study randomization, AND
  * Participant has no residual neurological dysfunction and has been off corticosteroids for at least 24 hours prior to sub-study randomization
* Participants must not have other known actionable oncogenic alterations, such as (but not limited to) EGFR sensitizing mutations, EGFR T790M mutation, ALK gene fusion, ROS1 gene rearrangement, RET gene rearrangement, NTRK rearrangement, HER2 mutation, KRAS activating mutations, and BRAF V600E mutation
* Participants who have received at least one line of systemic treatment for stage IV or recurrent NSCLC must have progressed (in the opinion of the treating physician) following the most recent line of therapy. Participants who have not yet received systemic treatment for their stage IV or recurrent NSCLC are allowed
* Participants may have received any number of lines of therapy for stage IV or recurrent NSCLC (including zero) and must be able to report prior treatment information
* Participants must have recovered (=< grade 1) from any side effects of prior therapy for NSCLC except alopecia and vitiligo
* Participants must not have received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) within 21 days prior to sub-study randomization
* Participants must not have received treatment with prior MET inhibitor therapies (e.g., crizotinib, tivantinib, savolitinib, tepotinib, cabozantinib, and foretinib).
* Participants must not have received treatment with prior angiogenesis inhibitor therapies (including but not limited to bevacizumab and ramucirumab)
* Participants must not have a history of interstitial lung disease that required steroid treatment
* Participants must not have received any radiation therapy within 7 days prior to sub-study randomization with the exceptions of

  * Stereotactic radiation to CNS metastases which must have been completed at least 3 days prior to sub-study randomization and
  * Palliative radiotherapy to bone metastases which must have been completed at least 1 day prior to sub-study randomization
* Participants must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study
* Participants must not have had a major surgery within 14 days prior to sub-study randomization. Participants must have fully recovered from the effects of prior surgery in the opinion of the treating investigator
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Absolute neutrophil count >= 1.5 x 10^3/uL (within 28 days prior to sub-study randomization)
* Hemoglobin >= 9.0 g/dL (within 28 days prior to sub-study randomization)
* Platelets >= 100 x 10^3/uL (within 28 days prior to sub-study randomization)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin =< 5 x institutional ULN (within 28 days prior to sub-study randomization)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 × institutional ULN. Participants with history of liver metastasis must have AST and ALT =< 5 x ULN (within 28 days prior to sub-study randomization)
* Participants must have a serum creatinine =< the institutional upper limit of normal (IULN) or calculated creatinine clearance >= 30 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to sub-study randomization
* Participants must have a cystatin C test performed to obtain baseline value within 28 days prior to sub-study randomization
* Participants' most recent Zubrod performance status must be 0-1 and be documented within 28 days prior to sub-study randomization
* Participants must have a completed medical history and physical exam within 28 days prior to sub-study randomization
* Participants must have adequate cardiac function. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy and have undetectable viral load test on the most recent test results obtained within 6 months prior to sub-study randomization
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to sub-study randomization, if indicated by the treating investigator
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to sub-study randomization, if indicated by the treating investigator
* Participants must not have cirrhosis at a level of Child-Pugh B (or worse) OR any degree of cirrhosis AND a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis
* Participants must not have grade < 0 of peripheral edema within 28 days prior to sub-study randomization
* Participants must not have experienced any arterial thromboembolic events, including but not limited to transient ischemic attack or cerebrovascular accident within 6 months prior to sub-study randomization
* Participants must not have uncontrolled blood pressure and hypertension within 28 days prior to sub-study randomization
* Participants must not be pregnant or breastfeeding (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must also be offered participation in specimen banking. With participant consent, specimens must be collected and submitted via the SWOG Specimen Tracking System
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines

  * NOTE: Participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Min Age: 18 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | Up to 3 years from date of sub-study randomization
  Rates will be compared using a chi-squared test at the 1-sided 10% level and also presented as the difference in response rates with the associated 80% confidence interval for the difference, Further, response rates and associated 80% confidence interval will be estimated for each arm.

SECONDARY OUTCOMES:
Incidence of treatment-related peripheral edema | Up to 3 years from date of sub-study randomization
  The frequency of peripheral edema will be compared using a 2-sided 10% level test of proportions. All-grade peripheral edema will be estimated along with 90% confidence intervals. Data from lymphoscintigraphy imaging will be summarized for baseline and among those with peripheral edema.
Incidence and severity of toxicities | Up to 3 years from date of sub-study randomization
  Toxicities combining the treatment arms and within each treatment arm will be reported.
Progression-free survival | From date of sub-study randomization to date of first documentation of progression or death due to any cause, assessed up to 3 years
  Will be estimated using the method of Kaplan-Meier. Will be compared between the arms using a 1-sided 10% level log-rank test. Medians and associated 80% confidence intervals will be estimated using the Brookmeyer-Crowley method.
Overall survival | Up to 3 years from date of sub-study randomization
  Will be estimated using the method of Kaplan-Meier. Medians and associated 80% confidence intervals will be estimated using the Brookmeyer-Crowley method.
Duration of response | From date of first documentation of response (complete response [CR] or partial response [PR]) to date of first documentation of progression or death due to any cause among participants who achieve a response (CR or PR), assessed up to 3 years
  Will be estimated using the method of Kaplan-Meier. Medians and associated 80% confidence intervals will be estimated using the Brookmeyer-Crowley method.

OTHER OUTCOMES:
Establishment of a tissue/blood repository | Up to 3 years from date of sub-study randomization

CONTACTS AND LOCATIONS:
Overall Officials: Paul K Paik, Principal Investigator — SWOG Cancer Research Network
Locations (267):
- United States (267):
  - Gulf Health Hospitals Inc/Infirmary Cancer Care - Malbis, Daphne, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Gulf Health Hospitals Inc/Infirmary Cancer Care - Saraland, Saraland, Alabama
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente Lutherville - Timonium Medical Center, Lutherville, Maryland
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Kaiser Permanente-Caton Hill Medical Center, Woodbridge, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin